CLINICAL TRIAL: NCT01847820
Title: Clinical Evaluation of the AmniSure ROM Test
Status: Terminated | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C13-ROM-001
Record Dates: First submitted 2013-05-01; First posted 2013-05-07 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Rupture of Fetal Membranes
Keywords: ROM; PROM; PPROM (preterm premature rupture of membranes)
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic: Individuals with signs, symptoms or suspicion of membrane rupture at 11 to 42 weeks gestation that will receive the AmniSure ROM test.
  Interventions: Device: AmniSure ROM test

INTERVENTIONS:
Device: AmniSure ROM test — Comparison of AmniSure ROM test to clinical diagnosis of ROM.

SUMMARY:
To show that having less qualified personnel (non-Laboratory trained professionals) perform the test yields the same result as if a Laboratory trained professional performed the test.

DETAILED DESCRIPTION:
The main goal of this study is to show that when performed by less qualified personnel, the AmniSure® ROM Test is so simple and accurate that the likelihood of erroneous results by the Intended-User is negligible and that the test poses no unreasonable risk of harm to the patient if performed incorrectly.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be pregnant.
* Subjects must be between 18 and 50 years of age and have a gestational age of 11.0-42.0 weeks.
* Subjects reporting suspicion, signs, or symptoms suggestive of ROM, PROM, PPROM.
* Subjects providing informed consent.

Exclusion Criteria:

* Subjects who have placenta previa.
* Subjects who have heavy vaginal bleeding.
* Subjects who have had digital vaginal examination immediately prior to evaluation for ROM.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be women presenting with signs, symptoms or suspicion of membrane rupture at 11 to 42 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The evaluation the clinical performance of the AmniSure® ROM test performed by the Intended-User relative to the clinical diagnosis of rupture of membranes. | One time at time of enrollment
  The investigational AmniSure ROM test will be compared to the three standard tests of nitrazine, ferning and pooling to determine rupture of fetal membranes.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco- Fresno, Fresno, California
  - Indiana University, Indianapolis, Indiana
  - Kansas University Medical Center Research Institute, Inc, Kansas City, Kansas
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Johnson JW, Daikoku NH, Niebyl JR, Johnson TR Jr, Khouzami VA, Witter FR. Premature rupture of the membranes and prolonged latency. Obstet Gynecol. 1981 May;57(5):547-56. PMID 7219903
- [Background] LEBHERZ TB, HELLMAN LP, MADDING R, ANCTIL A, ARJE SL. DOUBLE-BLIND STUDY OF PREMATURE RUPTURE OF THE MEMBRANES. A REPORT OF 1,896 CASES. Am J Obstet Gynecol. 1963 Sep 15;87:218-25. doi: 10.1016/0002-9378(63)90502-7. No abstract available. PMID 14077618
- [Background] Gunn GC, Mishell DR Jr, Morton DG. Premature rupture of the fetal membranes. A review. Am J Obstet Gynecol. 1970 Feb 1;106(3):469-83. doi: 10.1016/0002-9378(70)90378-9. No abstract available. PMID 4905833
- [Background] Sacks M, Baker TH. Spontaneous premature rupture of the membranes. A prospective study. Am J Obstet Gynecol. 1967 Apr 1;97(7):888-93. doi: 10.1016/0002-9378(67)90512-1. No abstract available. PMID 6021103
- [Background] Daikoku NH, Kaltreider DF, Khouzami VA, Spence M, Johnson JW. Premature rupture of membranes and spontaneous preterm labor: maternal endometritis risks. Obstet Gynecol. 1982 Jan;59(1):13-20. PMID 7078844
- [Background] Christensen KK, Christensen P, Ingemarsson I, Mardh PA, Nordenfelt E, Ripa T, Solum T, Svenningsen N. A study of complications in preterm deliveries after prolonged premature rupture of the membranes. Obstet Gynecol. 1976 Dec;48(6):670-7. PMID 825795
- [Background] Fayez JA, Hasan AA, Jonas HS, Miller GL. Management of premature rupture of the membranes. Obstet Gynecol. 1978 Jul;52(1):17-21. PMID 683624
- [Background] Alexander JM, Cox SM. Clinical course of premature rupture of the membranes. Semin Perinatol. 1996 Oct;20(5):369-74. doi: 10.1016/s0146-0005(96)80003-6. PMID 8912990
- [Background] Philipson EH, Hoffman DS, Hansen GO, Ingardia CJ. Preterm premature rupture of membranes: experience with latent periods in excess of seven days. Am J Perinatol. 1994 Nov;11(6):416-9. doi: 10.1055/s-2007-994609. PMID 7857433
- [Background] Lockwood CJ, Wein R, Chien D, Ghidini A, Alvarez M, Berkowitz RL. Fetal membrane rupture is associated with the presence of insulin-like growth factor-binding protein-1 in vaginal secretions. Am J Obstet Gynecol. 1994 Jul;171(1):146-50. doi: 10.1016/0002-9378(94)90461-8. PMID 7518190
- [Background] Fuks et al. N-Dia Amnisure Abstract.
- [Background] ACOG Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 80: premature rupture of membranes. Clinical management guidelines for obstetrician-gynecologists. Obstet Gynecol. 2007 Apr;109(4):1007-19. doi: 10.1097/01.AOG.0000263888.69178.1f. PMID 17400872
- [Background] Nisell H, Hagskog K, Westgren M. Assessment of fetal fibronectin in cervical secretion in cases of equivocal rupture of the membranes at term. Acta Obstet Gynecol Scand. 1996 Feb;75(2):132-4. doi: 10.3109/00016349609033304. PMID 8604598
- [Background] Atterbury JL, Groome LJ, Hoff C. Methods used to diagnose premature rupture of membranes: a national survey of 812 obstetric nurses. Obstet Gynecol. 1998 Sep;92(3):384-9. doi: 10.1016/s0029-7844(98)00178-1. PMID 9721775
- [Background] de Haan HH, Offermans PM, Smits F, Schouten HJ, Peeters LL. Value of the fern test to confirm or reject the diagnosis of ruptured membranes is modest in nonlaboring women presenting with nonspecific vaginal fluid loss. Am J Perinatol. 1994 Jan;11(1):46-50. doi: 10.1055/s-2007-994535. PMID 8155212
- [Background] Jeurgens-Borst AJ, Bekkers RL, Sporken JM, van den Berg PP. Use of insulin like growth factor binding protein-1 in the diagnosis of ruptured fetal membranes. Eur J Obstet Gynecol Reprod Biol. 2002 Apr 10;102(1):11-4. doi: 10.1016/s0301-2115(01)00560-7. PMID 12039083
- [Background] Watanabe T, Minakami H, Itoi H, Sato I, Sakata Y, Tamada T. Evaluation of latex agglutination test for alpha-fetoprotein in diagnosing rupture of fetal membranes. Gynecol Obstet Invest. 1995;39(1):15-8. doi: 10.1159/000292368. PMID 7534254
- [Background] Fujimoto S, Kishida T, Sagawa T, Negishi H, Okuyama K, Hareyama H, Makinoda S. Clinical usefulness of the dye-injection method for diagnosing premature rupture of the membranes in equivocal cases. J Obstet Gynaecol (Tokyo 1995). 1995 Jun;21(3):215-20. doi: 10.1111/j.1447-0756.1995.tb01000.x. PMID 8590356
- [Background] Birkenmaier A, Ries JJ, Kuhle J, Burki N, Lapaire O, Hosli I. Placental alpha-microglobulin-1 to detect uncertain rupture of membranes in a European cohort of pregnancies. Arch Gynecol Obstet. 2012 Jan;285(1):21-5. doi: 10.1007/s00404-011-1895-9. Epub 2011 Apr 8. PMID 21475966
- [Background] Lee SE, Park JS, Norwitz ER, Kim KW, Park HS, Jun JK. Measurement of placental alpha-microglobulin-1 in cervicovaginal discharge to diagnose rupture of membranes. Obstet Gynecol. 2007 Mar;109(3):634-40. doi: 10.1097/01.AOG.0000252706.46734.0a. PMID 17329514
- [Background] Eriksen NL, Parisi VM, Daoust S, Flamm B, Garite TJ, Cox SM. Fetal fibronectin: a method for detecting the presence of amniotic fluid. Obstet Gynecol. 1992 Sep;80(3 Pt 1):451-4. PMID 1495705
- [Background] El-Messidi A, Cameron A. Diagnosis of premature rupture of membranes: inspiration from the past and insights for the future. J Obstet Gynaecol Can. 2010 Jun;32(6):561-569. doi: 10.1016/S1701-2163(16)34525-X. PMID 20569537
- [Background] Hellemans P, Verdonk P, Baekelandt M, Joostens M, Francx M, Gerris J. Preliminary results with the use of the ROM-check immunoassay in the early detection of rupture of the amniotic membranes. Eur J Obstet Gynecol Reprod Biol. 1992 Feb 28;43(3):173-9. doi: 10.1016/0028-2243(92)90170-4. PMID 1563568
- [Background] Duff P & Lockwood, C. Diagnosis of Premature Rupture of Membranes.Up-to-Date, 2011.
- [Background] Di Renzo GC, Roura LC, Facchinetti F, Antsaklis A, Breborowicz G, Gratacos E, Husslein P, Lamont R, Mikhailov A, Montenegro N, Radunovic N, Robson M, Robson SC, Sen C, Shennan A, Stamatian F, Ville Y. Guidelines for the management of spontaneous preterm labor: identification of spontaneous preterm labor, diagnosis of preterm premature rupture of membranes, and preventive tools for preterm birth. J Matern Fetal Neonatal Med. 2011 May;24(5):659-67. doi: 10.3109/14767058.2011.553694. Epub 2011 Mar 2. No abstract available. PMID 21366393
- [Background] Sayres W. Chapter D: Preterm Labor & Premature Rupture of Membranes, AAFP-ALSO, June 2011.
- [Background] Mercer B. Premature Rupture of the Membranes. In: Gabbe SG, Niebyl JR, Galn HL, Jauniaux EM, Landon MB, Simpson JL, Driscoll DA, eds. Obstetrics: Normal and Problem Pregnancies. 6th ed. Philadelphia, PA: Saunders-Elsevier; 2012: 663.
- [Background] Mariona FG, Cabero L. Are we ready for a new look at the diagnosis of premature rupture of membranes? J Matern Fetal Neonatal Med. 2012 Apr;25(4):403-7. doi: 10.3109/14767058.2011.581715. Epub 2011 Jun 1. PMID 21627549
- [Background] Kurdoglu M, Kolusari A, Adali E, Yildizhan R, Kurdoglu Z, Kucukaydin Z, Kaya A, Kirimi E, Sahin HG, Kamaci M. Does residual amniotic fluid after preterm premature rupture of membranes have an effect on perinatal outcomes? 12 years experience of a tertiary care center. Arch Gynecol Obstet. 2010 Apr;281(4):601-7. doi: 10.1007/s00404-009-1147-4. Epub 2009 Jun 12. PMID 19521709
- [Background] Gungorduk K, Asicioglu O, Besimoglu B, Gungorduk OC, Yildirm G, Ark C, Sahbaz A. Labor induction in term premature rupture of membranes: comparison between oxytocin and dinoprostone followed 6 hours later by oxytocin. Am J Obstet Gynecol. 2012 Jan;206(1):60.e1-8. doi: 10.1016/j.ajog.2011.07.035. Epub 2011 Jul 30. PMID 21924396
- [Background] Combs CA, Garite TJ, Maurel K, Mallory K, Edwards RK, Lu G, Porreco R, Das A; Obstetrix Collaborative Research Network. 17-Hydroxyprogesterone caproate to prolong pregnancy after preterm rupture of the membranes: early termination of a double-blind, randomized clinical trial. BMC Res Notes. 2011 Dec 29;4:568. doi: 10.1186/1756-0500-4-568. PMID 22206581
- [Background] Derbent AU, Simavli SA, Kafali H, Turhan N. A comparison of subgroups of spontaneous preterm delivery: preterm labor with intact membranes and preterm premature rupture of membranes. Anatol J Obstet Gynecol 2012; 1: 1